CLINICAL TRIAL: NCT04375566
Title: Improving Decision Making by Developing and Testing a Progressive Web App About Patient Decision Aid for Stage I-II Non-small Cell Lung Cancer
Brief Title: Progressive Web App About Individualized Patient Decision Aid for NSCLC Stage I-II
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Other Study IDs: UM_iPDA_PM
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Lung Cancer Stage I; Lung Cancer Stage II
Keywords: iPDA; Shared decision making; Patient decision aids; Progressive web app
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- IT specialist: 20 IT Specialist will evaluate the usability and patient-friendliness of the tool
  Interventions: Other: Patient Decision Aid
- Doctors: 13 doctors will evaluate the information in the tool
  Interventions: Other: Patient Decision Aid
- Patients: 10-20 patients will evaluate the utility and the contribution of the tool in decision making proces.
  Interventions: Other: Patient Decision Aid

INTERVENTIONS:
Other: Patient Decision Aid — More than 20 IT specialists, 15 doctors and 15 patients

SUMMARY:
Studies indicate that the majority of early-stage non-small cell lung cancer (NSCLC) patients find it important to be involved in treatment decision making. However, in a recent study it has been reported that about 40% of the participants experienced decision conflict and feel uninformed(1). The investigators therefore developed a patient decision aid (PDA) for stage I-II NSCLC patients, that informs and empowers patients to help decide between stereotactic radiotherapy (SBRT) and surgery.

DETAILED DESCRIPTION:
A pilot study in which semi-structured interviews will be conducted (Qualitative research).In addition, patients will be asked to fill in a questionnaire about the usability of the prototype. A small group of patients (n=15) that have been treated for early stage NSCLC in the past will be asked to participate. The persons involved in this pilot are asked to assess a patient decision tool and will be interviewed only once. After the interview they will be asked to fill in a questionnaire. The burden of the pilot study is very low. No medical examinations or procedures will be carried out. Pilot study in lung cancer patients treated in the past with radiotherapy or surgery. The participants will all give informed consent. The investigators are using a qualitative design. Semi-structured interviews will be carried out. In addition the investigators will ask the participants to fill in a questionnaire with 35 questions.

No age limits are defined. The pilot study will be carried out in stage I-II NSCLC patients who were treated with radiotherapy or surgery, at least 6 months ago. Patients should currently be free of disease, no disease progression. The semi-structured interview consists of 17 open questions and text recorded, in order to be able to analyze the date afterwards. The interviews will take place when the patients come to the hospital for a regular follow-up appointment. After the interview, the patient is asked to fill in a questionnaire about the usability of the decision aid. In total, the expected duration is about 2 hours.

ELIGIBILITY:
Inclusion Criteria:

Early stage non-small cell lung patients, Treated with curative intent minimum 6 month ago, max 5 years. Doctors IT

Exclusion Criteria:

Others

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Included early stage lung cancer patients and doctors. 10-20 doctors 15 patients More than 20 IT specialists
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2021-10-04 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Usability of PDA | 1 year
  Opinion of the respondents about patient decision aid
The accuracy of the information in the tool | 1 year
  Testing the information provided in the tool and the usability of the tool itself

CONTACTS AND LOCATIONS:
Locations (1):
- Iva Halilaj, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No